CLINICAL TRIAL: NCT00520819
Title: Dietary Antioxidant Intervention in Smoking Middle-Aged and Elderly Men
Brief Title: Oslo Antioxidant Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Ullevaal University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OAS
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2007-08-27 (Estimated); Status verified 2007-08

CONDITIONS: Cardiovascular Disease
Keywords: Antioxidants; Phytochemicals; Oxidative stress; Inflammation; Endothelial function
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Antioxidant-rich food items

SUMMARY:
The primary objective of this study is to test whether increasing the total intake of antioxidants to middle-aged smoking men increases the antioxidant defence, reduces oxidative damage, and improves biomarkers for oxidative stress.

The secondary objectives is to test whether this strategy improves other cardiovascular risk markers including platelet function, lipid levels, inflammation, and markers of endothelial damage.

DETAILED DESCRIPTION:
In this study men smoking 5 or more cigarettes daily will be invited to participate. We will only include individuals with high cardiovascular risk (men rather than women, smokers rather than nonsmokers, middle-aged to elderly rather than young individuals), in order to recruit people with presumed high oxidative stress who might be most likely to show an effect and benefit from our intervention.

at the time of inclusion, participants will be randomized to three groups; control group, kiwi group or phytochemical group. The kiwi group will consume three kiwis a day, whereas the phytochemical group will consume an array of antioxidant-rich food stuffs. The intervention period is eight weeks.

Blood samples will be collected before and after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 45-75 years
* Daily smoker of a minimum of 5 cigarettes a day
* BMI <35 kg/m2 (because of difficulties that may be experienced by morbidly obese individuals in following the diet)
* Stable weight range of 4 kg or less during the previous 12 weeks

Exclusion Criteria:

* Any symptomatic CVD (myocardial infarction, angina pectoris, CABG, PCI, CHF, NYHA class III-IV)
* Diabetes type I or type II taking drugs for diabetes
* Following a vegetarian diet or near-vegetarian diet currently
* Allergy to nuts, kiwi fruits, chocolate, strawberries or tomatoes
* Clinical disorders including gastrointestinal disease impairing compliance with dietary recommendations
* History of serious or unstable medical or psychiatric disorder
* Current use of or need of lipid lowering drug treatment, aspirin or non-steroidal anti-inflammatory drugs (NSAID), according to assessment of the primary clinical investigator. Any "over the counter" headache/ pain or cold remedies taken during the study must not contain aspirin or aspirin like drugs such as ibuprofen. These are classed as and will interfere with platelet function, making them unresponsive for a period of 10-14 days. Paracetamol, however, can be taken as an alternative if required
* History of alcohol/or drug abuse
* Participation in a drug trial during the previous 30 days
* Use of drugs (Xenical, Reductil), nutritional supplements or herbs for weight loss within the 4 weeks prior to visit 2 or participation in an active weight reduction program
* Use of single vitamin or other antioxidants (must be stopped 4 weeks prior to visit 2)
* Individuals judged by the clinical investigator to be unable to follow instructions and procedures of the study.

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2003-02; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Biomarkers cardiovascular risk including platelet function, lipid levels, inflammation, and markers of endothelial damage. | 8 weeks

SECONDARY OUTCOMES:
Biomarkers cardiovascular risk including platelet function, lipid levels, inflammation, and markers of endothelial damage. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rune Blomhoff, PhD, Principal Investigator — University of Oslo; Serena Tonstad, MD, Principal Investigator — Ullevaal University Hospital; Anette Karlsen, MSc, Principal Investigator — University of Oslo
Locations (1):
- Ullevål University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Karlsen A, Svendsen M, Seljeflot I, Sommernes MA, Sexton J, Brevik A, Erlund I, Serafini M, Bastani N, Remberg SF, Borge GI, Carlsen MH, Bohn SK, Myhrstad MC, Dragsted LO, Duttaroy AK, Haffner K, Laake P, Drevon CA, Arnesen H, Collins A, Tonstad S, Blomhoff R. Compliance, tolerability and safety of two antioxidant-rich diets: a randomised controlled trial in male smokers. Br J Nutr. 2011 Aug;106(4):557-71. doi: 10.1017/S0007114511000353. PMID 21806852
- [Derived] Bohn SK, Myhrstad MC, Thoresen M, Holden M, Karlsen A, Tunheim SH, Erlund I, Svendsen M, Seljeflot I, Moskaug JO, Duttaroy AK, Laake P, Arnesen H, Tonstad S, Collins A, Drevon CA, Blomhoff R. Blood cell gene expression associated with cellular stress defense is modulated by antioxidant-rich food in a randomised controlled clinical trial of male smokers. BMC Med. 2010 Sep 16;8:54. doi: 10.1186/1741-7015-8-54. PMID 20846424